CLINICAL TRIAL: NCT03462927
Title: A Randomised, Open-label, Maximal Use Trial, Evaluating the Pharmacokinetic Profile of Active Ingredients and Their Metabolites After Application of MC2-01 Cream Compared With Active Comparator in Subjects With Extensive Psoriasis Vulgaris
Brief Title: A Maximal Use Trial Evaluating the Pharmacokinetic Profile of MC2-01 Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC2-01-C3
Record Dates: First submitted 2018-02-20; First posted 2018-03-13 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MC2-01 Cream (Experimental): MC2-01 cream (CAL and BDP, w/w 0.005%/ 0.064%).
  Interventions: Drug: MC2-01 Cream
- CAL/BDP combination (Active Comparator): CAL/BDP ointment (w/w 0.005%/0.064%).
  Interventions: Drug: CAL/BDP combination

INTERVENTIONS:
Drug: MC2-01 Cream — MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%)
  Arms: MC2-01 Cream
Drug: CAL/BDP combination — Calcipotriene/betamethasone (calcipotriene/ betamethasone dipropionate, w/w 0.005%/0.064%)
  Arms: CAL/BDP combination

SUMMARY:
This is a phase 2, randomised, open-label, parallel-group, multicentre trial in which MC2-01 cream and calcipotriene [CAL]/betamethasone [BDP] ointment (comparator) is investigated in subjects with clinically diagnosed extensive psoriasis vulgaris.

DETAILED DESCRIPTION:
The MC2-01 cream is designed for optimal patient satisfaction - it quickly absorbs into the skin leaving it nicely moisturized allowing patients to move on with daily routines. In this trial, the MC2-01 cream will be compared to a marketed calcipotriene [CAL]/betamethasone dipropionate [BDP] ointment. The purpose of the trial, is to determine the pharmacokinetic parameters of MC2-01 cream and the comparator under maximum use conditions.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent.
* Generally healthy males or non-pregnant females, of any race or ethnicity, who are at least 18 years of age at the time of screening.
* At Visit 1/Day 0, have a clinical diagnosis of plaque psoriasis (psoriasis vulgaris) of at least 6 months duration involving scalp and body (trunk and/or limbs) that is amenable to topical treatment with a maximum of 100 g of trial medication per week.
* Have a Physician's Global Assessment [PGA] of severity of at least moderate on the trunk, limbs and/or scalp, at Visit 1/Day 0.
* Have a treatment area between 20% and 30% of the body surface area [BSA] on the trunk, limbs and/or scalp, excluding psoriatic lesions on the face, genitals, and intertriginous areas, at Visit 1/Day 0.

Exclusion Criteria:

* Current diagnosis of unstable forms of psoriasis
* Other inflammatory skin disease in the treatment area
* Pigmentation, extensive scarring, pigmented lesions or sunburn in the treatment areas
* Planned exposure to natural or artificial sunlight
* Phototherapy and ultraviolet B radiation within 4 weeks prior to Visit 1/Baseline and during the trial;
* Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders;
* Oral calcium supplements, vitamin D supplements, bisphosphonates or calcitonin within 4 weeks prior to Visit 1/Day 0 during the trial period.
* Planned initiation of, or changes to concomitant medication that could affect calcium metabolism during the trial;
* Planned initiation of, or changes to, concomitant estrogen therapy during the trial;
* Strong systemic cytochrome P450 3A4 (CYP 3A4) inhibitors within 4 weeks prior to Vist 1/Day 0 and during the trial period;
* Use of topical treatments, except for emollients and non-medicated shampoos, with a possible effect on psoriasis within 2 weeks prior to Visit 1/Day 0 and during the trial period;
* Systemic treatment with biological therapies
* Initiation of, or expected changes to, concomitant medication that may affect psoriasis during the trial period;
* Depression and endocrine disorders known to affect cortisol levels or HPA axis integrity, non-nocturnal sleep patterns
* Systemic medication that suppresses the immune system within 4 weeks prior to the Visit 1/Day 0 and during the trial period;
* Clinical signs of skin infection with bacteria, viruses, or fungi;
* Known human immunodeficiency virus [HIV] infection;
* Known or suspected of hypersensitivity to any component of the test product or reference product;
* Any chronic or acute medical condition that may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-08-04 (Actual); Study Completion 2018-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Han, Principal Investigator — Department of Dermatology, Mount Sinai Beth Israel
Locations (1):
- Lenus Research and Medical Group, Sweetwater, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 08Feb-2018. Last Subject Last Visit: 04-Aug-2018.
Pre-assignment Details: Prior to randomization, the subject entered a washout period (if required) where anti-psoriatic treatment and other relevant medication/treatments were discontinued as defined by the exclusion criteria. The washout/screening period lasted for up to 4 weeks depending on which disallowed treatments the subject received.
Groups:
- MC2-01 Cream: MC2-01 cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/ 0.064%). One application daily for 8 weeks.
  MC2-01 Cream: MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%)
- CAL/BDP Combination: CAL/BDP ointment (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%, w/w 0.005%/0.064%). One daily application for 4 weeks.
  CAL/BDP combination: Calcipotriene/betamethasone (calcipotriene/ betamethasone dipropionate, w/w 0.005%/0.064%)
Period: Overall Study
Arm/Group | MC2-01 Cream | CAL/BDP Combination
Started | 32 | 31
Completed | 26 | 29
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.5) | 49.7 (16.2) | 51.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63
Baseline Physician's Global Assessment (PGA) [Count of Participants; unit: Participants] — Severity of psoriasis at Baseline
  Participants
    Moderate | 29 | 30 | 59
    Severe | 3 | 1 | 4
Baseline Body Surface Area (BSA) [Mean (Standard Deviation); unit: Percentage of psoriasis involvement] — Percentage involvement of psoriasis on the BSA at Baseline
  Percentage of psoriasis involvement | 23.56 (2.52) | 24.09 (3.13) | 23.82 (2.82)
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Measure Description: Fitzpatrick Skin Type was recorded at baseline using the following classification: I = Pale white skin, blue/hazel eyes, blond/red hair; II = Fair skin, blue eyes; III = Darker white skin; IV = Light brown skin; V = Brown skin; VI = Dark brown or black skin
  Participants
    I | 3 | 2 | 5
    II | 11 | 9 | 20
    III | 8 | 6 | 14
    IV | 5 | 9 | 14
    V | 3 | 5 | 8
    VI | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of the Active Ingredient Calcipotriene
Description: Geometric Mean for Maximum Plasma Concentration [Cmax] for the active ingredient Calcipotriene. Plasma concentration was measured at the following timepoints: pre-dose, 30 min, 1, 2, 3, 5 and 7 hours post-dose
Time Frame: Week 4
Population: 9 subjects were excluded from the PK evaluation at Week 4: 5 in the MC2-01 cream group and 4 in the active comparator group
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- MC2-01 Cream: MC2-01 cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%).
- CAL/BDP Ointment: CAL/BDP ointment: Calcipotriene/betamethasone (calcipotriene/ betamethasone dipropionate, w/w 0.005%/0.064%)
Arm/Group | MC2-01 Cream | CAL/BDP Ointment
Number analyzed (Participants) | 27 | 27
pg/mL | 30.2 [29.8 to 30.7] | 30.0 [30 to 30]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of the Active Ingredient Calcipotriene
Description: as for outcome 1
Time Frame: Week 8
Population: As per protocol, only subjects assigned to the MC2-01 cream had samples for PK testing collected at week 8. Only subjects that had a computable value of the PK parameter have been included in the analysis
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 19
pg/mL | 30.0 [30.0 to 30.0]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Active Ingredient Betamethasone Dipropionate
Description: Geometric Mean for Maximum Plasma Concentration [Cmax] for the active ingredient Betamethasone Dipropionate. Plasma concentration was measured at the following timepoints: pre-dose, 30 min, 1, 2, 3, 5 and 7 hours post-dose
Time Frame: Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- CAL/BDP Combination: CAL/BDP ointment: Calcipotriene/betamethasone (calcipotriene/ betamethasone dipropionate, w/w 0.005%/0.064%)
Arm/Group | MC2-01 Cream | CAL/BDP Combination
Number analyzed (Participants) | 27 | 27
pg/mL | 21.5 [19.5 to 23.7] | 23.1 [19.0 to 28.1]

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Active Ingredient Betamethasone Dipropionate
Description: as for outcome 3
Time Frame: Week 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 19
pg/mL | 20.0 [20.0 to 20.0]

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of the Metabolite MC1080
Description: Geometric Mean for Maximum Plasma Concentration [Cmax] for the metabolite MC1080. Plasma concentration was measured at the following timepoints: pre-dose, 30 min, 1, 2, 3, 5 and 7 hours post-dose
Time Frame: Week 4
Population: 9 subjects were excluded from the PK evaluation at Week 4: 5 in the MC2-01 cream group and 4 in active comparator group
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MC2-01 Cream | CAL/BDP Ointment
Number analyzed (Participants) | 27 | 27
pg/mL | 29.8 [28.7 to 31.0] | 29.2 [29.0 to 29.3]

6. Primary Outcome: Maximum Plasma Concentration (Cmax) of the Metabolite MC1080
Description: as for outcome 5
Time Frame: Week 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 19
pg/mL | 29.1 [29.1 to 29.1]

7. Primary Outcome: Maximum Plasma Concentration (Cmax) of Metabolite Betamethasone 17-propionate
Description: Geometric Mean for Maximum Plasma Concentration [Cmax] for the metabolite Betamethasone 17-propionate. Plasma concentration was measured at the following timepoints: pre-dose, 30 min, 1, 2, 3, 5 and 7 hours post-dose
Time Frame: Week 4
Population: 9 subjects were excluded from the PK evaluation at Week 4: 5 in the MC2-01 cream group and 4 in active comparator group
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MC2-01 Cream | CAL/BDP Ointment
Number analyzed (Participants) | 27 | 27
pg/mL | 39.3 [25.8 to 59.8] | 38.2 [27.4 to 53.4]

8. Primary Outcome: Maximum Plasma Concentration (Cmax) of Metabolite Betamethasone 17-propionate
Description: as for outcome 7
Time Frame: Week 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 19
pg/mL | 26.2 [20.5 to 33.5]

9. Secondary Outcome: Number of Subjects With Hypothalamic-pituitary-adrenal [HPA] Suppression After 4 Weeks of Treatment
Description: The HPA axis evaluation is based on an Adrenocorticotropic hormone [ACTH] challenge test, defined by a 30 minutes ACTH stimulated cortisol value. Only subject with no HPA suppression at baseline were included in the analysis.
  The outcome measure lists the number of subjects with HPA suppression 30 minutes after ACTH challenge
Time Frame: Week 4
Population: The HPA challenge test were only performed on subjects that were assigned to the MC2-01 cream group. No data were collected from the CAL/BDP Ointment group. Out of a total of 32 subjects, 5 subjects were excluded from the analysis as they had HPA suppression at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 27
Participants | 1

10. Secondary Outcome: Number of Subjects With Hypothalamic-pituitary-adrenal [HPA] Suppression After 8 Weeks of Treatment
Description: The HPA challenge test were only performed on subjects that were assigned to the MC2-01 cream group. Out of a total of 32 subjects, 5 subjects were excluded from the analysis as they had HPA suppression at baseline
Time Frame: Week 8
Population: The HPA challenge test were only performed on subjects that were assigned to the MC2-01 cream group. No data were collected from the CAL/BDP Ointment group. Out of a total of 32 subjects, 6 subjects were excluded from the analysis; 5 as they had HPA suppression at baseline and 1 who withdrew consent
Measure: Count of Participants; unit: Participants
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 26
Participants | 2

11. Secondary Outcome: Calcium Metabolism Evaluation in Albumin-corrected Serum Calcium
Description: Changes from baseline of albumin-corrected serum calcium [mmol/L]
Time Frame: Baseline and week 4
Population: As per protocol, only subjects assigned to the MC2-01 cream were included in the calcium metabolism evaluation. No data were collected from the CAL/BDP Ointment group. 5 subjects in the MC2-01 cream group were excluded from the analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 27
mmol/L | -0.00 (0.09)

12. Secondary Outcome: Calcium Metabolism Evaluation in Albumin-corrected Serum Calcium
Description: Changes from baseline in albumin-corrected serum calcium [mmol/L]
Time Frame: Baseline and week 8
Population: As per protocol, only subjects assigned to the MC2-01 cream were included in the calcium metabolism evaluation. No data were collected from the CAL/BDP Ointment group. 6 subjects in the MC2-01 cream group were excluded from the analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 26
mmol/L | 0.00 (0.07)

13. Secondary Outcome: Calcium Metabolism Evaluation of 24-hour Urinary Calcium Excretion
Description: Changes from baseline of 24-hour urinary calcium excretion [mmol/day]
Time Frame: Baseline and week 4
Population: As per protocol, only subjects assigned to the MC2-01 cream were included in the calcium metabolism evaluation. No data were collected from the CAL/BDP Ointment group. 8 subjects in the MC2-01 cream group were excluded from the analysis
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 24
mmol/day | -0.56 (1.69)

14. Secondary Outcome: Calcium Metabolism Evaluation of 24-hour Urinary Calcium Excretion
Description: Changes from baseline of 24-hour urinary calcium excretion [mmol/day]
Time Frame: Baseline and week 8
Population: As per protocol, only subjects assigned to the MC2-01 cream were included in the calcium metabolism evaluation. No data were collected from the CAL/BDP Ointment group. 12 subjects in the MC2-01 cream group were excluded from the analysis
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 20
mmol/day | -0.45 (1.08)

15. Secondary Outcome: Calcium Metabolism Evaluation of the Ratio of Urinary Calcium to Creatinine
Description: Changes from baseline in ratio of urinary calcium to creatinine defined as urinary calcium (mmol)/creatinine (g)
Time Frame: Baseline and week 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 24
mmol/g | -0.23 (1.49)

16. Secondary Outcome: Calcium Metabolism Evaluation of the Ratio of Urinary Calcium to Creatinine
Description: Changes from baseline in ratio of urinary calcium to creatinine defined as urinary calcium (mmol)/creatinine (g)
Time Frame: Baseline and week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 20
mmol/g | 0.00 (1.32)

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed from the time of the signature of the informed consent form by the subject during the screening visit (up to 4 weeks prior to treatment), during the treatment period (up to 8 weeks) and until the final follow-up visit had occurred (up to 4 weeks following end of treatment). All AEs that were considered related to the trial product would be followed until they were resolved, or until the medical condition of the subject was stable
Arm/Group | MC2-01 Cream | CAL/BDP Combination
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-01 Cream (N=32) | CAL/BDP Combination (N=31)
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT03462927/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03462927/SAP_001.pdf